CLINICAL TRIAL: NCT04914221
Title: A Randomized, Open-label, Single-dose, Replicate Crossover Study to Compare the Pharmacokinetics and Safety in Healthy Adult Volunteers Following Oral Administration of JLP-2002
Brief Title: The Safety and PK Characteristics of the Co-administration of JLP-2002 and Comparator in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jeil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: JLP-2002-101-PK
Record Dates: First submitted 2021-05-31; First posted 2021-06-04 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Overactive Bladder(OAB)
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (Experimental): Period I- comparator / Period II- comparator / Period III-JLP-2002
  Interventions: Drug: JLP-2002; Drug: Comparator
- Group II (Experimental): Period I- comparator / Period II- -JLP-2002 / Period III- comparator
  Interventions: Drug: JLP-2002; Drug: Comparator
- Group III (Experimental): Period I- JLP-2002/ Period II- comparator / Period III- comparator
  Interventions: Drug: JLP-2002; Drug: Comparator

INTERVENTIONS:
Drug: JLP-2002 — administration of JLP-2002
Drug: Comparator — administration of comparator

SUMMARY:
A randomized, open-label, single-dose, replicate crossover study to compare the pharmacokinetics and safety in healthy adult volunteers following oral administration of JLP-2002

DETAILED DESCRIPTION:
A randomized, open-label, single-dose, replicate crossover study

ELIGIBILITY:
Inclusion Criteria:

* Those who are 19 years of age or older and 55 years of age
* BMI 18.5 ~ 27.5 kg/m2
* Those who voluntarily agrees in writing after hearing a sufficient explanation of the purpose and procedure of the clinical trial

Exclusion Criteria:

* Those with clinically significant diseases or a history of liver, kidney, cardiovascular system, endocrine system, musculoskeletal system, respiratory system, neuropsychiatric system, blood/oncology system, etc.
* Those with a history of gastrointestinal diseases or surgery that may affect the absorption of drugs
* Those who donated whole blood within 60 days from the date of eligibility assessment, or who donated component blood within 30 days
* Those who do not have a medically recognized contraceptive intention or plan to provide sperm from the screening date to 4 weeks from the last administration of the investigational drug
* Those whose blood AST, ALT, or GGT levels in the screening test exceeded 3 times the upper limit of the reference range
* Those who showed clinically significant results in the hepatitis B test, hepatitis C test, HIV test, and syphilis test
* In the case of women, those who do not show a negative response on the pregnancy test
* Those who judged that the investigator is not suitable for participation in clinical trials, such as showing clinically significant results in other screening tests

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2021-03-13 (Actual); Primary Completion 2021-05-26 (Actual); Study Completion 2021-05-26 (Actual)

PRIMARY OUTCOMES:
AUClast of JLP-2002 | Time Frame: 192 hours
Cmax of JLP-2002 | Time Frame: 192 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea